CLINICAL TRIAL: NCT07381127
Title: A Study to Evaluate the Safety and Efficacy of Ionic Fluid in Treating Symptoms in Patients With Benign Prostatic Hyperplasia. A Prospective, Single-arm, Single-center Clinical Study.
Brief Title: INTUPRO in the Treatment of Benign Prostatic Hyperplasia-Related Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: inTumo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTUMO-003
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: BPH (Benign Prostatic Hyperplasia); BPH; BPH With Other Lower Urinary Tract Symptoms
Keywords: procedure; needle; benign prostate hyperplasia; moderate sedation; outpatient
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Under TRUS guidance, a fixed dose of the ablative agent will be administered to patients. Each patient will receive a total of 4-10 mL of ionic fluid, administered as two separate 2-5 mL injections into each side of the prostatic urethra.
  Interventions: Device: INTUPRO ionic fluid

INTERVENTIONS:
Device: INTUPRO ionic fluid — Under TRUS imaging, a fixed dose of the ablative agent will be administered to patients by the physician via needle. Each patient will receive a total of 4-10 mL ionic fluid , administered as two separate 2-5 mL injections into each side of the prostatic urethra.

SUMMARY:
The goal of this clinical trial is to determine whether INTUPRO can improve the quality of life in patients with Benign Prostate Hyperplasia (BPH).

The main questions it aims to answer are:

Can INTUPRO treatment lead to the removal of the Foley catheter? Can INTUPRO treatment improve urinary flow? Can INTUPRO treatment lower or minimize waking during sleep to urinate? Can INTUPRO reduce urinary hesitancy, urgency and frequency?

Participants will:

Receive INTUPRO treatment on Day 1. Visit at Day 30 and Day 90 for checkups, tests and Prostate MRI.

DETAILED DESCRIPTION:
The main goal of this study is to determine how well INTUPRO improves urinary symptoms in patients with benign prostatic hyperplasia (BPH). Effectiveness will be measured by changes in the International Prostate Symptom Score (IPSS), a standard questionnaire used to assess urinary symptoms.

Another goal of this study is to evaluate the safety of INTUPRO. This includes monitoring and recording all side effects, complications, or other medical problems that occur during the procedure and during the follow-up period after treatment.

This study is planned to last approximately one year; each patient will be followed for 3 months after treatment. Enrollment of 30 patients is expected.

ELIGIBILITY:
Inclusion Criteria:

* • Male patient aged 45 years or older

  * Prostate volume greater than 30 grams
  * An International Prostate Symptom Score (IPSS) of 12 or higher
  * Presence of obstructive urinary symptoms, such as difficulty starting urination, leakage of urine after voiding, or a feeling of incomplete bladder emptying.

This criterion may include patients who have previously been diagnosed with prostate cancer and completed treatment, but are experiencing urinary problems.

* Life expectancy of at least 3 months
* Ability to understand the study information and provide written informed consent
* Willingness and ability to comply with all study requirements, including procedures, clinical assessments, and follow-up visits

Exclusion Criteria:

* Urethral stricture

  * Bladder stones
  * Prostate volume 120 grams or greater
  * Presence of a prostate median lobe
  * History of bladder cancer or kidney cancer, and/or prior surgery related to these conditions
  * Previous radiation therapy to the pelvic region
  * Prior invasive surgical treatment for BPH symptoms
  * The Principal Investigator believes the patient would not tolerate the procedure
  * Presence of a cognitive impairment that, in the opinion of the Principal Investigator, would interfere with the patient's ability to provide reliable data or to safely complete the study
  * Bleeding disorders
  * Known allergy or intolerance to MRI contrast agents required for imaging used to evaluate treatment effectiveness after ionic fluid application
  * Other significant concurrent medical conditions that, in the investigator's judgment, could prevent clinical benefit from the procedure or could place the patient or study objectives at risk (including, but not limited to, active infection, kidney dysfunction, or significant comorbidities)
  * Significant medical or psychiatric illness
  * Participation in another clinical study involving a device, drug, or procedure that has not been completed or that could affect the outcomes of this study
  * Inability or unwillingness to undergo MRI examinations during the study period for any reason

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Urinary Symptoms (IPSS Score) | 3 months
  The change in the International Prostate Symptom Score (IPSS) from baseline will be evaluated after treatment. IPSS scores recorded at the screening visit will be compared with scores obtained at the 1-month and 3-month follow-up visits. A reduction in the IPSS score at 1 month and 3 months compared with baseline will be considered a primary outcome measure.
Procedure-Related and Post-Procedure Complications | 3 months
  Complications related to the procedure and the postoperative period will be assessed at 1 day, 1 month, and 3 months after treatment. The following complications will be specifically monitored:
  * Urinary retention
  * Urinary tract infection, suggested by a positive urine culture
  * Urosepsis
  * Blood in the urine (hematuria)
  * Perineal hematoma

SECONDARY OUTCOMES:
Procedure-Related Pain (Wong-Baker Pain Scale) | 3 months
  Pain related to the procedure will be assessed using the Wong-Baker Pain Scale on the day of treatment (Day 1), and at the 1-month and 3-month follow-up visits. Pain scores at follow-up visits will be compared with the pain level recorded on the day of the procedure.
Urinary Incontinence Symptoms (ICIQ-UI) | 3 months
  Changes in urinary incontinence symptoms will be evaluated using the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF). Scores will be recorded at baseline, 1 month, and 3 months after treatment, and follow-up scores will be compared with baseline values.
Sexual Function (IIEF Score) | 3 months
  Changes in erectile function will be assessed using the International Index of Erectile Function (IIEF). Scores will be collected at baseline, 1 month, and 3 months, and compared with baseline measurements.
Retrograde Ejaculation | 3 months
  The proportion of patients reporting retrograde ejaculation after the procedure will be recorded at the 1-month and 3-month follow-up visits.
Quality of Life Related to Urinary Symptoms (IPSS-QoL) | 3 months
  Changes in quality of life related to urinary symptoms will be assessed using the IPSS Quality of Life (IPSS-QoL) score. Measurements will be taken at baseline, 1 month, and 3 months, and follow-up scores will be compared with baseline values.
Uroflowmetry | 3 months
  Uroflowmetry measurements (Qmax - maximum flow rate, mL/s) will be collected at the 1-month and 3-month follow-up visits and compared with baseline values.
Pressure-Flow Study (If Performed) | 3 months
  In patients who undergo pressure-flow studies, Detrusor pressure at Qmax (Pdet@Qmax) will be recorded at baseline and, if available, at the 1-month and 3-month follow-up visits, and compared with baseline values.
Presence of prostate tissue ablation | 3 months
  The presence and extent of prostate tissue ablation (complete, partial, none) will be evaluated using MRI (or other imaging methods, if applied) at baseline, 1 month, and 3 months. Imaging findings will be compared across time points.
Post-Procedure Urinary Catheterization Time | 3 months
  The total duration of urinary catheter use after the procedure, measured in days, will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital Research Center, Istanbul, Turkey (Türkiye)